CLINICAL TRIAL: NCT00361959
Title: Multicentre, Randomised, Double-Blind, Double Dummy, Parallel Group, 104-week Study to Compare the Effect of the Salmeterol/Fluticasone Propionate Combination Product (SERETIDE*) 50/500mcg Delivered Twice Daily Via the DISKUS*/ACCUHALER* Inhaler With Tiotropium Bromide 18 mcg Delivered Once Daily Via the HandiHaler Inhalation Device on the Rate of Health Care Utilisation Exacerbations in Subjects With Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: SERETIDE 50/500mcg Versus Tiotropium Bromide On Exacerbation Rates In Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO40036
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: fluticasone propionate/salmeterol combination; tiotropium; SERETIDE; COPD exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Fluticasone

INTERVENTIONS:
Drug: Tiotropium bromide 18mcg
Drug: Fluticasone propionate/ salmeterol combination 50/500mcg
  Other Names: Tiotropium bromide 18mcg

SUMMARY:
This is a comparator study to assess the relative efficacy of the combination product fluticasone propionate/salmeterol 50/500 and tiotropium bromide on the rate of exacerbations of chronic obstructive pulmonary disease (COPD) over a two year study interval.

DETAILED DESCRIPTION:
A Multicentre, Randomised, Double-Blind, Double Dummy, Parallel Group, 104 Week Study to Compare the Effect of the Salmeterol/Fluticasone Propionate Combination Product (SERETIDE) 50/500mcg with Tiotropium Bromide 18 mcg on the Rate of Exacerbations in Subjects with Severe Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion criteria:

* Established clinical history of moderate to severe COPD.
* Post bronchodilator FEV1 of < 50% of predicted normal.
* FEV1 / FVC ratio <70%.
* Reversibility to 400mcg albuterol of less or equal to 10 predicted at Visit 1.
* Free from exacerbation in the 6 weeks prior to screening.
* Current or former smoker with a smoking history of = 10 pack-years and has a history of COPD exacerbations.

Exclusion criteria:

* Current asthma, eczema, atopic dermatitis and/or allergic rhinitis.
* Has a known respiratory disorder other than COPD (e.g. lung cancer, sarcoidosis, tuberculosis or lung fibrosis).
* Has narrow-angle glaucoma, prostatic hyperplasia or obstruction of the neck of the bladder that in the opinion of the investigator should prevent the subject from entering the study.
* Has undergone lung transplantation and/or lung volume reduction.
* Female who is a nursing mother.
* Requires regular (daily) long-term oxygen therapy (LTOT).
* Is receiving beta-blockers (except eye drops).
* Has a serious, uncontrolled disease likely to interfere with the study.
* Has received any other investigational drugs within the 4 weeks prior to Visit 1.
* Has, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse.
* Has a known or suspected hypersensitivity to beta2-agonists, inhaled corticosteroids, anticholinergic agents or any components of the formulations (e.g. lactose or milk protein).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1270 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Rate of healthcare utilisation based exacerbations of COPD

SECONDARY OUTCOMES:
Rates for exacerbations based on symptoms, treatment with oral corticosteroids and for antibioticsTime to next exacerbation, duration and difference between healthcare utilisation and symptom based exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (135):
- Austria (4):
  - GSK Investigational Site, Grimmenstein
  - GSK Investigational Site, Mödling
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Belgium (6):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Czechia (6):
  - GSK Investigational Site, Blansko
  - GSK Investigational Site, Kyjov
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Odense C
- Estonia (4):
  - GSK Investigational Site, Paide
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (13):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bad Kissingen, Bavaria
  - GSK Investigational Site, Bad Tölz, Bavaria
  - GSK Investigational Site, Bad Woerrishofen, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (6):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Chania, Crete
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Kavala
  - GSK Investigational Site, Periohi Dragana, Alexandroupolis
  - GSK Investigational Site, Rethymnon, Crete
- Italy (15):
  - GSK Investigational Site, Cassano Murge (BA), Apulia
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Eboli (SA), Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, Telese (BN), Campania
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rivolta d'Adda (CR), Lombardy
  - GSK Investigational Site, Sesto San Giovanni (MI), Lombardy
  - GSK Investigational Site, Ascoli Piceno, The Marches
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, San Sisto (PG), Umbria
  - GSK Investigational Site, Padua, Veneto
- Latvia (2):
  - GSK Investigational Site, Jēkabpils
  - GSK Investigational Site, Riga
- Lithuania (4):
  - GSK Investigational Site, Alytus
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Netherlands (18):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Leiderdorp
  - GSK Investigational Site, Meppel
  - GSK Investigational Site, Oss
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Venlo
  - GSK Investigational Site, Weert
  - GSK Investigational Site, Zwolle
- Norway (9):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Egsjordet
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Gjettum
  - GSK Investigational Site, Moelv
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Trondheim
  - GSK Investigational Site, Tønsberg
  - GSK Investigational Site, Volda
- Romania (4):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
- Russia (3):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Slovakia (4):
  - GSK Investigational Site, Bardejov
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Prievidza
- Slovenia (4):
  - GSK Investigational Site, Golnik
  - GSK Investigational Site, Litija
  - GSK Investigational Site, Topolšica
  - GSK Investigational Site, Zgornje Hoče
- Spain (9):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Figueres
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Orihuela (Alicante)
  - GSK Investigational Site, Vic
  - GSK Investigational Site, Zaragoza
- Sweden (8):
  - GSK Investigational Site, Eksjö
  - GSK Investigational Site, Karlstad
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Ukraine (2):
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
- United Kingdom (9):
  - GSK Investigational Site, Peterborough, Cambridgeshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Liverpool, Lancashire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Isleworth, Middlesex
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, Birmingham, Warwickshire
  - GSK Investigational Site, London
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Calverley PMA, Stockley RA, Seemungal TAR, Hagan G, Willits LR, Riley JH, Wedzicha JA; Investigating New Standards for Prophylaxis in Reduction of Exacerbations (INSPIRE) Investigators. Reported pneumonia in patients with COPD: findings from the INSPIRE study. Chest. 2011 Mar;139(3):505-512. doi: 10.1378/chest.09-2992. Epub 2010 Jun 24. PMID 20576732
- [Background] Chui D, Tejani AM. The INSPIRE trial results: are they truly breathtaking? Am J Respir Crit Care Med. 2009 Jan 1;179(1):80; author reply 80-1. doi: 10.1164/ajrccm.179.1.80. No abstract available. PMID 19098157
- [Background] Hilleman DE, Malesker MA, Morrow LE, Schuller D. A systematic review of the cardiovascular risk of inhaled anticholinergics in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2009;4:253-63. doi: 10.2147/copd.s4620. Epub 2009 Jul 20. PMID 19657399
- [Background] Lanes SF, Jara M. The INSPIRE study: influence of prior use and discontinuation of inhaled corticosteroids. Am J Respir Crit Care Med. 2008 Sep 1;178(5):543-4; author reply 544. doi: 10.1164/ajrccm.178.5.543. No abstract available. PMID 18713851
- [Background] Middleton PG. Management of patients with COPD: a comparison of the INSPIRE and TORCH studies. Am J Respir Crit Care Med. 2008 Jul 1;178(1):106; author reply 106-7. doi: 10.1164/ajrccm.178.1.106. No abstract available. PMID 18565964
- [Background] Wedzicha JA, Calverley PM, Seemungal TA, Hagan G, Ansari Z, Stockley RA; INSPIRE Investigators. The prevention of chronic obstructive pulmonary disease exacerbations by salmeterol/fluticasone propionate or tiotropium bromide. Am J Respir Crit Care Med. 2008 Jan 1;177(1):19-26. doi: 10.1164/rccm.200707-973OC. Epub 2007 Oct 4. PMID 17916806
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: SCO40036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCO40036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCO40036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCO40036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCO40036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCO40036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCO40036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register